CLINICAL TRIAL: NCT02051218
Title: Prevention of Symptomatic Skeletal Events With Denosumab Administered Every 4 Weeks Versus Every 12 Weeks - A Non-Inferiority Phase III Trial
Brief Title: Prevention of Symptomatic Skeletal Events With Denosumab Administered Every 4 Weeks Versus Every 12 Weeks
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SAKK 96/12; 000000685 (Other: SNCTP); 2014-001189-87 (EudraCT Number)
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer; Metastatic Prostate Cancer; Bone Metastases
Keywords: metastatic breast cancer; castration resistant metastatic prostate cancer; bone metastases; Denosumab; XGEVA; de-escalation
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (standard arm) (Active Comparator): Denosumab 120mg (XGEVA®) sc. q4w
  Interventions: Drug: Denosumab (standard dosing)
- Arm B (reduced arm) (Experimental): Denosumab 120mg (XGEVA®) sc. q4w [weeks 1, 5, 9] followed by Denosumab 120mg (XGEVA®) sc. q12w [weeks 13, 25, …]
  Interventions: Drug: Denosumab (reduced dosing)

INTERVENTIONS:
Drug: Denosumab (reduced dosing) — 3x Denosumab 120mg (XGEVA®) sc. q4w followed by Denosumab 120mg (XGEVA®) sc. q12w
  Other Names: XGEVA®
  Arms: Arm B (reduced arm)
Drug: Denosumab (standard dosing) — Denosumab 120mg (XGEVA®) sc. q4w
  Other Names: XGEVA®
  Arms: Arm A (standard arm)

SUMMARY:
The aim of the trial is to test the hypothesis that the benefit of denosumab is maintained if administered only every 12 weeks as compared to every 4 weeks.

DETAILED DESCRIPTION:
Denosumab, a monoclonal antibody against RANK-Ligand has been shown superior to zoledronic acid in delaying time to a first on-study skeletal related event (SRE) in patients with solid tumors, with no effects on disease progression or survival. Many SREs were silent compression fractures found only because of scheduled imaging. The approved dose of denosumab is 120 mg s.c. every 4 weeks (q4w). Although generally well tolerated, there is a time-dependent increase in osteonecrosis of the jaw in up to 8% of patients. Cases of fatal hypocalcaemia were observed during post marketing surveillance.

The optimal dose and schedule for denosumab is unknown. Denosumab is associated with considerable costs and may add toxicity; thus a study of de-escalation is warranted.

The aim of the trial is to test the hypothesis that the benefit of Denosumab is maintained if administered 120 mg q12w as compared to 120 mg q4w. The primary endpoint of this open-label randomized phase III non-inferiority trial is time to first on-trial symptomatic skeletal event (SSE: i.e. clinically significant pathological fracture, radiation therapy to bone, surgery to bone or spinal cord compression). With a non-inferiority margin of 1.2 for the hazard ratio, a power 80% and a type I error 5%, the total sample size is 1380. Secondary endpoints are safety, time to subsequent on-trial SSE, quality of life, health economic outcomes, and change in bone turnover markers. This study is open for international collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent.
* Histologically confirmed diagnosis of breast or prostate cancer before randomization.
* Patient has metastatic breast cancer (stage IV, all subtypes allowed) or prostate cancer (stage IV) and bone metastases and is planned to receive or is receiving antineoplastic treatment.
* Patients with prostate cancer must have evidence of disease progression on continuous androgen deprivation therapy (CRPC).
* Patients must have ≥ 3 bone metastases (lytic or blastic or mixed). The lesions must be documented by radiological evaluation within 12 weeks before randomization (by X-Ray, CT scan, PET-CT, MRI scan or bone scintigraphy).
* WHO performance status 0-2
* Age ≥ 18 years.
* Corrected serum calcium ≥ 2 mmol/l and ≤ 3 mmol/l (medical treatments to obtain serum calcium levels in the normal range are allowed, as far as no denosumab is used. Maximally 1 dose of bisphosphonates in the case of hypercalcemia is allowed, if the bisphosphonate was applied at least 3 weeks before the first dose of denosumab).
* Liver transaminases not more than 1.5 x ULN or not more than 3 x ULN with liver metastases. Serum total bilirubin ≤ 1.5 x ULN (≤ 2.0 x ULN in case of known Gilbert's disease)
* Women are not breastfeeding. Women with child-bearing potential are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and during the 12 months thereafter. A negative pregnancy test before inclusion (within 7 days) into the trial is required for all women with child-bearing potential.
* Men agree not to father a child during participation in the trial and during 12 months thereafter.

Exclusion Criteria:

* Definite contraindication for denosumab (e.g. hypocalcaemia [Albumin-corrected serum calcium < 2.0 mmol/l]).
* History or current evidence of osteonecrosis of the jaw.
* Non-healed mucosa in oral cavity (by surgery or as a side effect of any other treatment).
* Jaw or dental conditions that require oral surgery or if surgery or invasive dental procedures are planned.
* Prior use of denosumab for bone metastases (dose 120 mg every 4 weeks) or bisphosphonates to treat bone metastases. Patients treated with denosumab or bisphosphonates against osteopenia or osteoporosis are allowed to enter the trial if the last dose was more than 28 days before randomization.
* Patients with known osteoporosis (T-score ≤ -2.5) at study entry (since fractures from osteoporosis are difficult to be discriminated from fractures through bone metastases).
* Radiotherapy or surgery to the bone within the last two weeks before randomization or planned within 6 weeks after randomization.
* Presence or history of CNS metastases or leptomeningeal disease. A MRI evaluation within 12 weeks before randomization must be performed in case of suspicious symptoms.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent, filling out QoL forms.
* Concurrent treatment in a clinical trial with SSE or SRE as primary endpoint.
* Known hypersensitivity to trial drug or hypersensitivity to any other component of the trial drug (e.g. fructose).
* Any concomitant drugs contraindicated for use with the trial drugs according to the approved product information.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the trial protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2014-07-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to first on-trial symptomatic skeletal event (SSE; Clinically significant pathological fracture, radiation therapy to bone, surgery to bone or spinal cord compression). | at the latest 5 years after randomization.
  A SSE is defined as one of the following events: Clinically significant pathological fracture, radiation therapy to bone, surgery to bone, or spinal cord compression.

SECONDARY OUTCOMES:
Toxicity (focus on hypocalcaemia and osteonecrosis of the jaw) | at the latest 5 years after randomization.
Time to first and subsequent on-trial SSE | at the latest 5 years after randomization.
Quality of Life measured by FACT-G and FACT-BP | at the latest 5 years after randomization.
Skeletal morbidity period rate (SMPR) | at the latest 5 years after randomization.
Skeletal morbidity rate (SMR) | at the latest 5 years after randomization.
Health economic analysis | at the latest 5 years after randomization.
Bone turnover markers | at the latest 5 years after randomization.
Overall Survival (OS) | at the latest 5 years after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Roger von Moos, PD MD, Study Chair — Kantonsspital Graubünden; Arnoud Templeton, MD, Study Chair — Cantonal Hospital of St. Gallen; Silke Gillessen, Prof, Study Chair — Cantonal Hospital of St. Gallen; Andreas Müller, MD, Study Chair — Kantonsspital Winterthur KSW
Locations (49):
- Austria (2):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Klinikum Wels-Grieskrichen GmbH, Wels
- Germany (5):
  - Uniklinik Düsseldorf, Urologische Klinik, Düsseldorf
  - Universitätsklinikum Düsseldorf, Frauenheilkunde/Geburtshilfe, Düsseldorf
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitäts-Frauenklinik Ulm, Ulm
- Switzerland (42):
  - Hirslanden Klinik Aarau, Aarau
  - Kantonspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - Brustzentrum Basel - Praxis für ambulante Tumortherapie, Basel
  - St. Claraspital AG, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Klinik Engeried / Praxis Oncocare, Bern
  - Inselspital, Bern, Bern
  - Spitalzentrum Biel, Biel
  - Spitalzentrum Oberwallis, Brig
  - Centre du Sein de Genève, Clinique des Grangettes, Chêne-Bougeries
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Frauenfeld - Brustzentrum, Frauenfeld
  - Hopital Fribourgeois, Fribourg
  - Hopitaux Universitaires de Geneve, Geneva
  - Clinique De Genolier, Genolier
  - Hôpital neuchâtelois, La Chaux-de-Fonds
  - CCAC Lausanne, Lausanne
  - CHUV, Lausanne
  - Kantonsspital Liestal, Liestal
  - Fondazione Oncologia / Oncologia ematologia, Locarno
  - Luzerner Kantonsspital, Lucerne
  - Hirslanden Klinik St. Anna Luzern, Lucerne
  - Oncologia Varini & Calderoni & Christinat, Lugano
  - Onkologie Zentrum Spital Männedorf, Männedorf
  - Kantonsspital Muensterlingen, Münsterlingen
  - Kantonsspital Olten, Olten
  - Tumor and Brustzentrum Ostschweiz TBZO, Sankt Gallen
  - Kantonsspital St. Gallen, Sankt Gallen
  - Rundum Onkologie am Bahnhofpark, Sargans
  - Spital Limmattal, Schlieren
  - Hôpital du Valais Sion, Sion
  - Bürgerspital Solothurn - Zentrum für Onkologie und Hämatologie, Solothurn
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Winterthur
  - Onkologie Bellevue, Zurich
  - Brustzentrum-Zürich, Zurich
  - Klinik für Hämatologie und Onkologie Hirslanden Zürich AG, Zurich
  - Onkozentrum Klinik im Park, Zurich
  - Universitätsspital Zürich, Zurich
  - Stadtspital Zürich Triemli, Zurich

REFERENCES:
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716